CLINICAL TRIAL: NCT03824106
Title: Frailty Rehabilitation: A Community-based Intervention to Promote Healthy Aging
Brief Title: Frailty Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 5500
Record Dates: First submitted 2019-01-22; First posted 2019-01-31 (Actual); Last update posted 2025-07-06 (Actual); Status verified 2024-11

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty | interventions — Nutritional Status; Medication Review; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm1.Control (Experimental): Participants randomized to the control arm will not receive any of the Frailty Rehabilitation Interventions. Participants in the control arm will receive Vitamin D.
  Interventions: Other: Control; Dietary Supplement: Vitamin D
- Arm2.Group Exercise (Experimental): Participants will attend the exercise program, twice-weekly, for 4-months with supplemental home exercise.
  Interventions: Behavioral: Group Exercise; Dietary Supplement: Vitamin D
- Arm3.Multi-modal Intervention (Experimental): Group Exercise/Supplemental Home Exercise: This will be delivered identically to Arm 2.
  Nutrition, protein supplementation, and a medication review will also be implemented.
  Interventions: Behavioral: Group Exercise; Combination Product: Nutrition and Medication review; Dietary Supplement: Protein Supplement; Dietary Supplement: Vitamin D

INTERVENTIONS:
Other: Control — Participants randomized to the control arm will not receive any of the Frailty Management Interventions.
  Arms: Arm1.Control
Behavioral: Group Exercise — A recent meta-analysis suggests 180 min/week of exercise (with a high challenge to balance) is most effective for fall prevention. Combined strength and endurance training performed at a moderate weekly frequency (i.e., two times per week) may promote marked gains on muscle hypertrophy, strength and power gains in frail older adults. Balance training is a key component of successful exercise programs for vulnerable older adults.
  Arms: Arm2.Group Exercise; Arm3.Multi-modal Intervention
Combination Product: Nutrition and Medication review — Nutrition review: Conduct nutritional screening flow and review any questions, provide some additional counseling/coaching. Protein supplements will be provided to all participants unless contraindicated.
  Medication review: Review/update current medication list and forward the list and medical history to the consultant study pharmacist.
  Arms: Arm3.Multi-modal Intervention
Dietary Supplement: Protein Supplement — Protein supplementation will be provided.
  Arms: Arm3.Multi-modal Intervention
Dietary Supplement: Vitamin D — 1000 IU of oral vitamin D

SUMMARY:
Frailty is an important clinical state that contributes to falls, hospitalization, institutionalization and death. When an individual simultaneously has many health problems, a frailty "tipping point" may be triggered by even a minor stressful event such as adding a new drug or urinary tract infection. Our research suggests that approximately 23% of Canadians over age 65 are frail, and by age 85 this estimate increases to over 40%. As we learn more about frailty and its consequences, there is an urgent need to develop community-based interventions that will prevent or delay frailty in older adults. Our proposed study will examine if frailty rehabilitation program is an effective community-based intervention to promote healthy aging. The primary objective of our study is to determine if 4-month frailty rehabilitation improves physical function compared with control and exercise alone in community-dwelling older adults living with frailty and sarcopenia. Secondary objectives of our study are to determine if 4-months of frailty rehabilitation can improve functional abilities and reduce healthcare utilization during a 6-month follow-up period compared with control and exercise alone. Results will translate the first Canadian model of frailty and sarcopenia rehabilitation and management.

DETAILED DESCRIPTION:
In this multi-arm randomized controlled trial (RCT), 324 community-dwelling older adults (aged 65+) with frailty and at high risk for mobility disability will be randomized into one of three arms (control, exercise only, multi-modal rehabilitation) stratified by sex, age and location preference. Rolling recruitment will occur with ten cohorts total (2-3 cohorts per site, n=33 participants per cohort), enrolled across the partner Young Men's Christian Association (YMCA) sites.

Building upon the RCT, we aim to understand which components of a functional rehabilitation program are essential to change the trajectory of sarcopenia in older adults and explore the feasibility of a functional rehabilitation program with older adults. All participants will be screened for sarcopenia at baseline. Of the 324 participants, a subset of participants with sarcopenia will undergo additional assessments.

A validated frailty questionnaire can be administered over the phone and will provide an estimate of frailty status.

Stratified block randomization (1:1 randomization ratio) with the allocation sequence generated by a computer will be used to randomly allocate eligible participants to their group assignment. Participants will be stratified based on their sex, age (<80 or >=80 years), and location preference. To protect against selection bias, the randomization sequence will be adequately concealed so that investigators/participants are not aware of the upcoming assignment. The proposed duration of treatment is 4-months.

Primary and secondary outcomes will be assessed at 0 and 4-months.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling ≥65 years of age
* Able to independently ambulate 25m with or without walking aid
* At high risk for mobility disability/functional limitations
* Received medical clearance
* Can arrange transportation to the YMCA up to 2x/week
* Proof of being fully vaccinated against COVID-19 and proof of identification

Exclusion Criteria:

* Unable to speak or understand English
* Currently attending a group exercise program
* Currently in a drug optimization study/program
* Currently taking protein supplements daily
* Significant cognitive impairment where they may have difficulty following two-step commands in group exercise
* Receiving palliative/end of life care
* Unstable angina or heart failure
* Unable to attend for more than 20% of trial duration

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Physical Performance | Baseline and 4-months
  Physical function will be assessed with the Short Performance Physical Battery [total score]. Higher scores indicate better physical performance [range 0-12].
Change in Walking Speed | Baseline and 4-months
  Walking speed will be assessed with the 400-m Walk Test [walking speed, m/s]. Faster walking speeds indicate better performance.

SECONDARY OUTCOMES:
Change in Frailty | Baseline and 4-months
  Frailty will be assessed with the Fit-Frailty App [total score]. Higher scores indicate greater frailty [range 0-1].
Change in Fear of Falling | Baseline and 4-months
  Iconographical Falls Efficacy Scale [total score]. Higher scores indicate greater fear of falling [range 16-28]
Change in Balance Confidence | Baseline and 4-months
  Dichotomous questions (y/n)
Change in Falls | Baseline and 4-months
  Number of falls will be assessed by self-report.
Change in Fitness | Baseline and 4-months
  Fitness will be assessed with Fitness Trackers [average step count per day]. A greater number of steps indicates higher fitness level.
Change in Strength | Baseline and 4-months
  Strength will be assessed with a handgrip dynamometer [kg].
Change in Functional Mobility | Baseline and 4-months
  Strength will be assessed with the Timed Up and Go (TUG) Test [total time]. A higher score indicates a greater falls risk (greater or equal to 12 sec) and lower functional mobility.
Change in Cognition | Baseline and 4-months
  Cognition will be assessed with the Montreal Cognitive Assessment [total score]. Higher scores indicate better cognition [range 0-30].
Change in Cognition | Baseline and 4-months
  Cognition will be assessed with the Mini-Mental State Examination [total score]. Higher scores indicate better cognition [range 0-30].
Change in Health-related Quality of Life | Baseline and 4-months
  Health-related quality of life will be assessed using a EuroQol instrument. Higher scores indicate better health-related quality of life [range 0-100].
Change in Life Space Mobility | Baseline and 4-months
  Life space mobility will be assessed with the Life Space Assessment [total score]. Higher scores indicate a larger life space [range 0-120].
Change in Basic Activities of Daily Living | Baseline and 4-months
  Activities of daily living will be assessed with the Katz activities of daily living questionnaire [total score]. Lower scores indicate greater impairment [range 0-6].
Change in Instrumental Activities of Daily Living | Baseline and 4-months
  Activities of daily living will be assessed with Lawton instrumental activities of daily living questionnaire [total scores]. Lower scores indicate greater impairment [range 0-8].
Change in Depression / Mood | Baseline and 4-months
  Depression and mood will be assessed with the Geriatric Depression Scale Short-Form [total score]. Higher scores indicate more depressive symptoms [range 0-15].
Change in Nutrition | Baseline and 4-months
  Nutrition will be assessed with the Mini Nutritional Assessment [total score]. Lower scores indicate malnutrition [range 0-14].
Change in Sarcopenia | Baseline and 4-months
  Sarcopenia will be assessed with the strength, assistance walking, rise from a chair, climb stairs, and falls (SARC-F) questionnaire [total score]. High scores (greater than or equal to 4) is predictive of sarcopenia [range 0-10].
Change in Muscle Mass | Baseline and 4-months
  Muscle mass will be assessed with dual-energy x-ray absorptiometry (DXA) and magnetic resonance imaging (MRI). A subset of participants will be assessed.
Change in Emergency Room Visits | Baseline, 4-months and additional 6-month follow-up
  Number of emergency room visits will be recorded. Higher number of emergency room visits indicates higher healthcare utilization.
Change in Hospitalizations | Baseline, 4-months and additional 6-month follow-up
  Number of hospitalizations will be recorded. Higher number of hospitalizations indicates higher healthcare utilization.
Change in Institutionalization | Baseline, 4-months and additional 6-month follow-up
  Institutionalization to long-term care will be recorded. Higher number individuals entering long-term care indicates higher healthcare utilization.

OTHER OUTCOMES:
Individual-level Economic Evaluation | Baseline, 4-months and additional 6-month follow-up
  Individual-level economic evaluations will be assessed by changes in direct medical costs and effectiveness outcomes (e.g., quality-adjusted life years - QALYs), calculate and compare the incremental cost-effectiveness ratio (ICER) (e.g., $/ QALY gained, $/ a visit averted) against a willingness-to-pay threshold ($50,000/QALY) to show if this program of frailty rehabilitation represents good value for money.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papaioannou, MD, MSc, Principal Investigator — McMaster University
Locations (1):
- McMaster University - St. Peter's Hospital, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Rockwood K, Mitnitski A. Frailty defined by deficit accumulation and geriatric medicine defined by frailty. Clin Geriatr Med. 2011 Feb;27(1):17-26. doi: 10.1016/j.cger.2010.08.008. PMID 21093719
- [Background] Kennedy CC, Ioannidis G, Rockwood K, Thabane L, Adachi JD, Kirkland S, Pickard LE, Papaioannou A. A Frailty Index predicts 10-year fracture risk in adults age 25 years and older: results from the Canadian Multicentre Osteoporosis Study (CaMos). Osteoporos Int. 2014 Dec;25(12):2825-32. doi: 10.1007/s00198-014-2828-9. Epub 2014 Aug 8. PMID 25103215
- [Background] Rockwood K, Song X, Mitnitski A. Changes in relative fitness and frailty across the adult lifespan: evidence from the Canadian National Population Health Survey. CMAJ. 2011 May 17;183(8):E487-94. doi: 10.1503/cmaj.101271. Epub 2011 Apr 26. PMID 21540166
- [Background] Roberts KC, Rao DP, Bennett TL, Loukine L, Jayaraman GC. Prevalence and patterns of chronic disease multimorbidity and associated determinants in Canada. Health Promot Chronic Dis Prev Can. 2015 Aug;35(6):87-94. doi: 10.24095/hpcdp.35.6.01. PMID 26302227
- [Background] Rockwood K, Howlett SE, MacKnight C, Beattie BL, Bergman H, Hebert R, Hogan DB, Wolfson C, McDowell I. Prevalence, attributes, and outcomes of fitness and frailty in community-dwelling older adults: report from the Canadian study of health and aging. J Gerontol A Biol Sci Med Sci. 2004 Dec;59(12):1310-7. doi: 10.1093/gerona/59.12.1310. PMID 15699531
- [Background] Cameron ID, Fairhall N, Langron C, Lockwood K, Monaghan N, Aggar C, Sherrington C, Lord SR, Kurrle SE. A multifactorial interdisciplinary intervention reduces frailty in older people: randomized trial. BMC Med. 2013 Mar 11;11:65. doi: 10.1186/1741-7015-11-65. PMID 23497404
- [Background] Morley JE, Vellas B, van Kan GA, Anker SD, Bauer JM, Bernabei R, Cesari M, Chumlea WC, Doehner W, Evans J, Fried LP, Guralnik JM, Katz PR, Malmstrom TK, McCarter RJ, Gutierrez Robledo LM, Rockwood K, von Haehling S, Vandewoude MF, Walston J. Frailty consensus: a call to action. J Am Med Dir Assoc. 2013 Jun;14(6):392-7. doi: 10.1016/j.jamda.2013.03.022. PMID 23764209
- [Background] Anderson L, Oldridge N, Thompson DR, Zwisler AD, Rees K, Martin N, Taylor RS. Exercise-Based Cardiac Rehabilitation for Coronary Heart Disease: Cochrane Systematic Review and Meta-Analysis. J Am Coll Cardiol. 2016 Jan 5;67(1):1-12. doi: 10.1016/j.jacc.2015.10.044. PMID 26764059
- [Background] Dalal HM, Doherty P, Taylor RS. Cardiac rehabilitation. BMJ. 2015 Sep 29;351:h5000. doi: 10.1136/bmj.h5000. No abstract available. PMID 26419744
- [Background] Cheifetz O, Park Dorsay J, Hladysh G, Macdermid J, Serediuk F, Woodhouse LJ. CanWell: meeting the psychosocial and exercise needs of cancer survivors by translating evidence into practice. Psychooncology. 2014 Feb;23(2):204-15. doi: 10.1002/pon.3389. Epub 2013 Sep 6. PMID 24009181
- [Background] Cheifetz O, Dorsay JP, MacDermid JC. Exercise facilitators and barriers following participation in a community-based exercise and education program for cancer survivors. J Exerc Rehabil. 2015 Feb 28;11(1):20-9. doi: 10.12965/jer.150183. eCollection 2015 Feb. PMID 25830140
- [Background] Theou O, Stathokostas L, Roland KP, Jakobi JM, Patterson C, Vandervoort AA, Jones GR. The effectiveness of exercise interventions for the management of frailty: a systematic review. J Aging Res. 2011 Apr 4;2011:569194. doi: 10.4061/2011/569194. PMID 21584244
- [Background] Sherrington C, Michaleff ZA, Fairhall N, Paul SS, Tiedemann A, Whitney J, Cumming RG, Herbert RD, Close JCT, Lord SR. Exercise to prevent falls in older adults: an updated systematic review and meta-analysis. Br J Sports Med. 2017 Dec;51(24):1750-1758. doi: 10.1136/bjsports-2016-096547. Epub 2016 Oct 4. PMID 27707740
- [Background] Fairhall N, Aggar C, Kurrle SE, Sherrington C, Lord S, Lockwood K, Monaghan N, Cameron ID. Frailty Intervention Trial (FIT). BMC Geriatr. 2008 Oct 13;8:27. doi: 10.1186/1471-2318-8-27. PMID 18851754
- [Background] Ng TP, Feng L, Nyunt MS, Feng L, Niti M, Tan BY, Chan G, Khoo SA, Chan SM, Yap P, Yap KB. Nutritional, Physical, Cognitive, and Combination Interventions and Frailty Reversal Among Older Adults: A Randomized Controlled Trial. Am J Med. 2015 Nov;128(11):1225-1236.e1. doi: 10.1016/j.amjmed.2015.06.017. Epub 2015 Jul 6. PMID 26159634
- [Background] Kelaiditi E, Cesari M, Canevelli M, van Kan GA, Ousset PJ, Gillette-Guyonnet S, Ritz P, Duveau F, Soto ME, Provencher V, Nourhashemi F, Salva A, Robert P, Andrieu S, Rolland Y, Touchon J, Fitten JL, Vellas B; IANA/IAGG. Cognitive frailty: rational and definition from an (I.A.N.A./I.A.G.G.) international consensus group. J Nutr Health Aging. 2013 Sep;17(9):726-34. doi: 10.1007/s12603-013-0367-2. PMID 24154642
- [Background] Negm AM, Kennedy CC, Thabane L, Veroniki AA, Adachi JD, Richardson J, Cameron ID, Giangregorio A, Papaioannou A. Management of frailty: a protocol of a network meta-analysis of randomized controlled trials. Syst Rev. 2017 Jul 5;6(1):130. doi: 10.1186/s13643-017-0522-7. PMID 28679416
- [Background] Haslam C, Cruwys T, Haslam SA. "The we's have it": evidence for the distinctive benefits of group engagement in enhancing cognitive health in aging. Soc Sci Med. 2014 Nov;120:57-66. doi: 10.1016/j.socscimed.2014.08.037. Epub 2014 Aug 28. PMID 25222136
- [Background] Papaioannou A, Kennedy CC, Giangregorio L, Ioannidis G, Pritchard J, Hanley DA, Farrauto L, DeBeer J, Adachi JD. A randomized controlled trial of vitamin D dosing strategies after acute hip fracture: no advantage of loading doses over daily supplementation. BMC Musculoskelet Disord. 2011 Jun 20;12:135. doi: 10.1186/1471-2474-12-135. PMID 21689448
- [Background] Visser M, Deeg DJ, Lips P; Longitudinal Aging Study Amsterdam. Low vitamin D and high parathyroid hormone levels as determinants of loss of muscle strength and muscle mass (sarcopenia): the Longitudinal Aging Study Amsterdam. J Clin Endocrinol Metab. 2003 Dec;88(12):5766-72. doi: 10.1210/jc.2003-030604. PMID 14671166
- [Background] Houston DK, Cesari M, Ferrucci L, Cherubini A, Maggio D, Bartali B, Johnson MA, Schwartz GG, Kritchevsky SB. Association between vitamin D status and physical performance: the InCHIANTI study. J Gerontol A Biol Sci Med Sci. 2007 Apr;62(4):440-6. doi: 10.1093/gerona/62.4.440. PMID 17452740
- [Background] Bruyere O, Cavalier E, Souberbielle JC, Bischoff-Ferrari HA, Beaudart C, Buckinx F, Reginster JY, Rizzoli R. Effects of vitamin D in the elderly population: current status and perspectives. Arch Public Health. 2014 Sep 28;72(1):32. doi: 10.1186/2049-3258-72-32. eCollection 2014. PMID 25279143
- [Background] Muir SW, Montero-Odasso M. Effect of vitamin D supplementation on muscle strength, gait and balance in older adults: a systematic review and meta-analysis. J Am Geriatr Soc. 2011 Dec;59(12):2291-300. doi: 10.1111/j.1532-5415.2011.03733.x. PMID 22188076
- [Background] Stockton KA, Mengersen K, Paratz JD, Kandiah D, Bennell KL. Effect of vitamin D supplementation on muscle strength: a systematic review and meta-analysis. Osteoporos Int. 2011 Mar;22(3):859-71. doi: 10.1007/s00198-010-1407-y. Epub 2010 Oct 6. PMID 20924748
- [Background] Halfon M, Phan O, Teta D. Vitamin D: a review on its effects on muscle strength, the risk of fall, and frailty. Biomed Res Int. 2015;2015:953241. doi: 10.1155/2015/953241. Epub 2015 Apr 27. PMID 26000306
- [Background] Cadore EL, Rodriguez-Manas L, Sinclair A, Izquierdo M. Effects of different exercise interventions on risk of falls, gait ability, and balance in physically frail older adults: a systematic review. Rejuvenation Res. 2013 Apr;16(2):105-14. doi: 10.1089/rej.2012.1397. PMID 23327448
- [Background] Kramer IF, Verdijk LB, Hamer HM, Verlaan S, Luiking YC, Kouw IWK, Senden JM, van Kranenburg J, Gijsen AP, Bierau J, Poeze M, van Loon LJC. Both basal and post-prandial muscle protein synthesis rates, following the ingestion of a leucine-enriched whey protein supplement, are not impaired in sarcopenic older males. Clin Nutr. 2017 Oct;36(5):1440-1449. doi: 10.1016/j.clnu.2016.09.023. Epub 2016 Sep 29. PMID 27743615
- [Background] Drey M, Pfeifer K, Sieber CC, Bauer JM. The Fried frailty criteria as inclusion criteria for a randomized controlled trial: personal experience and literature review. Gerontology. 2011;57(1):11-8. doi: 10.1159/000313433. Epub 2010 Apr 21. PMID 20407227
- [Background] Tieland M, van de Rest O, Dirks ML, van der Zwaluw N, Mensink M, van Loon LJ, de Groot LC. Protein supplementation improves physical performance in frail elderly people: a randomized, double-blind, placebo-controlled trial. J Am Med Dir Assoc. 2012 Oct;13(8):720-6. doi: 10.1016/j.jamda.2012.07.005. Epub 2012 Aug 11. PMID 22889730
- [Background] Kim CO, Lee KR. Preventive effect of protein-energy supplementation on the functional decline of frail older adults with low socioeconomic status: a community-based randomized controlled study. J Gerontol A Biol Sci Med Sci. 2013 Mar;68(3):309-16. doi: 10.1093/gerona/gls167. Epub 2012 Aug 9. PMID 22879453
- [Background] Cooper JA, Cadogan CA, Patterson SM, Kerse N, Bradley MC, Ryan C, Hughes CM. Interventions to improve the appropriate use of polypharmacy in older people: a Cochrane systematic review. BMJ Open. 2015 Dec 9;5(12):e009235. doi: 10.1136/bmjopen-2015-009235. PMID 26656020
- [Background] Page AT, Clifford RM, Potter K, Schwartz D, Etherton-Beer CD. The feasibility and effect of deprescribing in older adults on mortality and health: a systematic review and meta-analysis. Br J Clin Pharmacol. 2016 Sep;82(3):583-623. doi: 10.1111/bcp.12975. Epub 2016 Jun 13. PMID 27077231
- [Background] Hogan DB, Borrie M, Basran JF, Chung AM, Jarrett PG, Morais JA, Peters E, Rockwood KJ, St John PD, Sclater AL, Stultz T, Woolmore-Goodwin S. Specialist physicians in geriatrics-report of the canadian geriatrics society physician resource work group. Can Geriatr J. 2012 Sep;15(3):68-79. doi: 10.5770/cgj.15.41. Epub 2012 Sep 20. PMID 23259019
- [Background] Graham ID, Logan J, Harrison MB, Straus SE, Tetroe J, Caswell W, Robinson N. Lost in knowledge translation: time for a map? J Contin Educ Health Prof. 2006 Winter;26(1):13-24. doi: 10.1002/chp.47. PMID 16557505
- [Background] Bischoff-Ferrari HA, Dawson-Hughes B, Staehelin HB, Orav JE, Stuck AE, Theiler R, Wong JB, Egli A, Kiel DP, Henschkowski J. Fall prevention with supplemental and active forms of vitamin D: a meta-analysis of randomised controlled trials. BMJ. 2009 Oct 1;339:b3692. doi: 10.1136/bmj.b3692. PMID 19797342
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Rockwood K, Mitnitski A. Frailty in relation to the accumulation of deficits. J Gerontol A Biol Sci Med Sci. 2007 Jul;62(7):722-7. doi: 10.1093/gerona/62.7.722. PMID 17634318
- [Background] LIFE Study Investigators; Pahor M, Blair SN, Espeland M, Fielding R, Gill TM, Guralnik JM, Hadley EC, King AC, Kritchevsky SB, Maraldi C, Miller ME, Newman AB, Rejeski WJ, Romashkan S, Studenski S. Effects of a physical activity intervention on measures of physical performance: Results of the lifestyle interventions and independence for Elders Pilot (LIFE-P) study. J Gerontol A Biol Sci Med Sci. 2006 Nov;61(11):1157-65. doi: 10.1093/gerona/61.11.1157. PMID 17167156
- [Background] Fielding RA, Rejeski WJ, Blair S, Church T, Espeland MA, Gill TM, Guralnik JM, Hsu FC, Katula J, King AC, Kritchevsky SB, McDermott MM, Miller ME, Nayfield S, Newman AB, Williamson JD, Bonds D, Romashkan S, Hadley E, Pahor M; LIFE Research Group. The Lifestyle Interventions and Independence for Elders Study: design and methods. J Gerontol A Biol Sci Med Sci. 2011 Nov;66(11):1226-37. doi: 10.1093/gerona/glr123. Epub 2011 Aug 8. PMID 21825283
- [Background] Kwon S, Perera S, Pahor M, Katula JA, King AC, Groessl EJ, Studenski SA. What is a meaningful change in physical performance? Findings from a clinical trial in older adults (the LIFE-P study). J Nutr Health Aging. 2009 Jun;13(6):538-44. doi: 10.1007/s12603-009-0104-z. PMID 19536422
- [Background] Rockwood K, Andrew M, Mitnitski A. A comparison of two approaches to measuring frailty in elderly people. J Gerontol A Biol Sci Med Sci. 2007 Jul;62(7):738-43. doi: 10.1093/gerona/62.7.738. PMID 17634321
- [Background] Li G, Thabane L, Papaioannou A, Adachi JD. Comparison between frailty index of deficit accumulation and fracture risk assessment tool (FRAX) in prediction of risk of fractures. Bone. 2015 Aug;77:107-14. doi: 10.1016/j.bone.2015.04.028. Epub 2015 Apr 25. PMID 25916552
- [Background] Moore JB, Mitchell NG, Kilpatrick MW, Bartholomew JB. The physical self-attribute questionnaire: development and initial validation. Psychol Rep. 2007 Apr;100(2):627-42. doi: 10.2466/pr0.100.2.627-642. PMID 17564239
- [Background] Vasunilashorn S, Coppin AK, Patel KV, Lauretani F, Ferrucci L, Bandinelli S, Guralnik JM. Use of the Short Physical Performance Battery Score to predict loss of ability to walk 400 meters: analysis from the InCHIANTI study. J Gerontol A Biol Sci Med Sci. 2009 Feb;64(2):223-9. doi: 10.1093/gerona/gln022. Epub 2009 Jan 31. PMID 19182232
- [Background] Brach M, Moschny A, Bucker B, Klaassen-Mielke R, Trampisch M, Wilm S, Platen P, Hinrichs T. Recruiting hard-to-reach subjects for exercise interventions: a multi-centre and multi-stage approach targeting general practitioners and their community-dwelling and mobility-limited patients. Int J Environ Res Public Health. 2013 Dec 2;10(12):6611-29. doi: 10.3390/ijerph10126611. PMID 24317380
- [Background] McHenry JC, Insel KC, Einstein GO, Vidrine AN, Koerner KM, Morrow DG. Recruitment of Older Adults: Success May Be in the Details. Gerontologist. 2015 Oct;55(5):845-53. doi: 10.1093/geront/gns079. Epub 2012 Aug 16. PMID 22899424
- [Background] Dolovich L, Oliver D, Lamarche L, Agarwal G, Carr T, Chan D, Cleghorn L, Griffith L, Javadi D, Kastner M, Longaphy J, Mangin D, Papaioannou A, Ploeg J, Raina P, Richardson J, Risdon C, Santaguida PL, Straus S, Thabane L, Valaitis R, Price D. A protocol for a pragmatic randomized controlled trial using the Health Teams Advancing Patient Experience: Strengthening Quality (Health TAPESTRY) platform approach to promote person-focused primary healthcare for older adults. Implement Sci. 2016 Apr 5;11:49. doi: 10.1186/s13012-016-0407-5. PMID 27044360
- [Background] Kaczorowski J, Chambers LW, Karwalajtys T, Dolovich L, Farrell B, McDonough B, Sebaldt R, Levitt C, Hogg W, Thabane L, Tu K, Goeree R, Paterson JM, Shubair M, Gierman T, Sullivan S, Carter M. Cardiovascular Health Awareness Program (CHAP): a community cluster-randomised trial among elderly Canadians. Prev Med. 2008 Jun;46(6):537-44. doi: 10.1016/j.ypmed.2008.02.005. Epub 2008 Feb 14. PMID 18372036
- [Background] Kennedy CC, Thabane L, Ioannidis G, Adachi JD, Papaioannou A; ViDOS Investigators. Implementing a knowledge translation intervention in long-term care: feasibility results from the Vitamin D and Osteoporosis Study (ViDOS). J Am Med Dir Assoc. 2014 Dec;15(12):943-5. doi: 10.1016/j.jamda.2014.05.007. Epub 2014 Jun 18. PMID 24953541
- [Background] Kennedy CC, Ioannidis G, Giangregorio LM, Adachi JD, Thabane L, Morin SN, Crilly RG, Marr S, Josse RG, Lohfeld L, Pickard LE, King S, van der Horst ML, Campbell G, Stroud J, Dolovich L, Sawka AM, Jain R, Nash L, Papaioannou A. An interdisciplinary knowledge translation intervention in long-term care: study protocol for the vitamin D and osteoporosis study (ViDOS) pilot cluster randomized controlled trial. Implement Sci. 2012 May 24;7:48. doi: 10.1186/1748-5908-7-48. PMID 22624776
- [Background] Gafni A, Birch S. Incremental cost-effectiveness ratios (ICERs): the silence of the lambda. Soc Sci Med. 2006 May;62(9):2091-100. doi: 10.1016/j.socscimed.2005.10.023. Epub 2005 Dec 1. PMID 16325975